CLINICAL TRIAL: NCT01973088
Title: Screening and Identification of Human Urate Transporter hURAT1 MicroRNA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Qian-wei Li (Other)
Responsible Party: Sponsor-Investigator, Qian-wei Li, Southwest Hospital, China, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Other Study IDs: Southwest Hospital,TMMU
Record Dates: First submitted 2013-10-20; First posted 2013-10-31 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-09

CONDITIONS: Urinary Calculi
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- non-urate calculus
- non-calculus
- urate calculus

SUMMARY:
This study intends to use in patients with renal tissue and blood samples, screening and identification of renal tissue hURAT1 regulating the expression of micro-RNA, for further study of uric acid stone formation mechanism and the occurrence of clinical preventive uric acid stones provide new clues and new intervention targets.

ELIGIBILITY:
Inclusion Criteria:

A、B group were enrolled standards: ① aged 18-65 years old; ② comply with percutaneous nephrolithotomy lithotripsy indications for surgery; ③ ECT tips ipsilateral normal or mildly impaired renal function.

Group C patients were enrolled standards: ① aged 18-65 years old; ② normal renal function, not associated with urinary calculi in patients; ③ cancer patients met radical nephrectomy indications for surgery; ④ emergency trauma patients suffering from kidney resection surgical indications.

Exclusion Criteria:

* aged <18 years or> 65 years; ② neurological disease or cognitive dysfunction; ③ can not be corrected or uncorrected coagulopathy; ④ associated with diabetes, hypertension and other metabolic diseases; ⑤ accompanied by tuberculosis, hepatitis, HIV and other infectious diseases; ⑥ poor tolerance to anesthesia and surgery, such as: severe cardiopulmonary disease, coagulation disorders, etc.; ⑦ ultrasound, renal imaging examination revealed renal cortex was significantly thinner (renal cortical thickness <1.5cm), structural variation; ⑧ with severe systemic or urinary tract infection; ⑨ ECT tips ipsilateral renal function is severely impaired or solitary kidney.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Experiment are divided into uric acid stones group (A), non-uric acid stones group (B), control group (C), A, C recruited 30 patients each group, B group recruited 20 patients.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
micro-RNA | 6 months
  microRNA microarray:the micro-RNA of kidney tissue

SECONDARY OUTCOMES:
Urine | 24 hours
  Urine Analyzer:Urine color, transparency, pH, erythrocytes, leukocytes, epithelial cells, casts, protein, specific gravity, and qualitative urine
24h urine quantitative analysis | 96 hours
  Urine Analyzer:Urine, sodium, potassium, calcium, magnesium, ammonium, phosphate, sulfate, uric acid, oxalate, citrate, creatinine
Blood biochemistry | 24 hours
  Blood biochemical analyzer:Sodium, potassium, chloride, calcium, phosphorus, magnesium, bicarbonate, uric acid, creatinine
Stone analysis | 3 weeks
  Infrared Spectroscopy:Calcium oxalate monohydrate , carbonated apatite, calcium oxalate dihydrate ,anhydrous uric acid, urine ammonium,magnesium ammonium phosphate
hURAT1 transporter protein | 6 months
  WESTERN BLOT、RT-qPCR:hURAT1 transporter protein of kidney tissue